CLINICAL TRIAL: NCT00759642
Title: Phase II Trial of Lapatinib in Women With Hormone Receptor Positive (Estrogen Receptor [ER] and/or Progesterone Receptor [PR] +) Human Epidermal Growth Factor Receptor 2 (HER-2) Negative Metastatic Breast Cancer Who Have Failed Prior Antihormone Therapy
Brief Title: Lapatinib in Women With Metastatic Breast Cancer Who Have Failed Prior Antihormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB decision
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11495
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; hormone receptor positive; HER-2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib (Experimental): lapatinib
  Interventions: Drug: lapatinib

INTERVENTIONS:
Drug: lapatinib — lapatinib 1500 mg PO daily
  Other Names: Tykerb

SUMMARY:
Hormone receptor positive breast cancer is the most common type of breast cancer, comprising 70-80% of all breast cancers. Endocrine therapy is the main type of initial treatment for patients with your type of breast cancer. Endocrine therapy is treatment that tries to remove, or block certain hormones from binding to the cancer cells and thus slow or stop the growth of cancer. Although most patients with your type of breast cancer respond initially to endocrine therapies, it can lose its effectiveness. New therapies for this type of cancer are needed.

DETAILED DESCRIPTION:
Endocrine therapy forms the backbone of treatment for both early stage and advanced stage hormone receptor positive breast cancer. Although most patients with advanced estrogen receptor positive metastatic disease respond initially to endocrine therapies, this response is short lived. New therapies able to provide additional benefit to patients with hormone receptor positive, endocrine-resistant, advanced metastatic breast cancer are required. This study proposes to add lapatinib to endocrine therapy to treat hormone receptor positive HER-2 negative metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed invasive breast cancer, which at time of study entry is either stage III (locally advanced) disease not amenable to curative therapy or stage IV disease. Histological confirmation of recurrent/metastatic disease is encouraged but not required if clinical evidence of stage IV disease recurrence is available.
* ER and/or Progesterone Receptor (PgR )positive breast cancer (10% or more of infiltrating cancer cells exhibit nuclear staining for ER and/or PgR)
* Have had progressive disease or development of new metastatic disease while on treatment or within 12 months of treatment with an aromatase inhibitor and/or Fulvestrant in adjuvant or metastatic setting
* Have measurable (defined as at least 1 lesion that can be accurately measured in at least 1 dimension [longest diameter to be recorded], with minimum lesion size ≥ 2cm on conventional measurement techniques or ≥ 1cm on spiral computed tomography [CT] scan), or evaluable disease. Patients with lytic or blastic bone disease as only site of disease will be eligible for the study. These patients will be evaluable for progression but not for response.
* Primary tumor was HER-2 negative (IHC 0 or IHC 1+/2+ and Fluorescence in situ hybridization [FISH] ≤ 1.9)
* Patients could have received prior Tamoxifen either as adjuvant therapy or for stage IV disease
* Performance status of 2 or better per Eastern Cooperative Oncology Group (ECOG) criteria
* Adequate cardiac function (cardiac ejection fraction ≥ 50% as measured by echocardiogram or multigated acquisition (MUGA) scan).
* IV bisphosphonate and denosumab for bony metastatic disease will be allowed
* Palliative radiation therapy to bony metastases will be allowed
* Adequate bone marrow function per good medical practice. Results of these tests do not determine eligibility. Minor deviations are acceptable if they do not impact safety in the judgment of the treating physician. Absolute neutrophil count (ANC) ≥ 1500/mm3, platelet count ≥ 100,000/mm3, and hemoglobin ≥ 10 g/dL
* Adequate kidney function: serum creatinine of ≤ 1.5mg/dl and/or creatinine clearance of ≥ 60 mL/min
* Adequate hepatic function: transaminases < 2 x upper limit of normal and total bilirubin ≤ 1.5 mg/dL.
* Must have a serum albumin ≥ 3.0 g/dL.
* Must be informed of investigational nature of study and must sign informed consent in accordance with institutional rules.
* Pretreatment lab values must be performed within 14 days of patient registration and other baseline studies within 30 days.
* Patients will have a baseline bone scan, Computerized Tomography (CT) chest, abdomen and pelvis or Positron Emission Tomography (PET)/CT.
* If previously treated brain metastasis and free of central nervous system (CNS) symptoms and > 3 months from treatment of brain metastasis are eligible

Exclusion Criteria

* Prior HER-2 targeted therapy for metastatic disease
* Has uncontrolled brain metastasis or leptomeningeal disease
* Has rapidly progressing and/or bulky disease which in the opinion of the investigator may be more appropriately treated with a chemotherapy-based strategy.
* Has an uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring parenteral antibiotics or psychiatric illness/social situations that would limit compliance with study requirements.
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (eg, Crohn's, ulcerative colitis).
* Current active hepatic or biliary disease (exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Renal function as measured by creatinine clearance <3 0ml/min (ratio to norm < 0.1)
* HIV-positive patients receiving combination antiretroviral therapy
* Pregnant women
* Active cardiac disease defined as:

  * History of uncontrolled or symptomatic angina
  * History of arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation
  * Myocardial infarction < 6 months from study entry
  * Uncontrolled or symptomatic congestive heart failure
  * Ejection fraction below institutional normal limit
  * Any other cardiac condition, which in the opinion of treating physician, would make this protocol unreasonably hazardous for the patient
* History of another primary cancer, with exception of:

  * curatively resected nonmelanomatous skin cancer
  * curatively treated cervical carcinoma in-situ
  * other primary solid tumor curatively resected treated with no known active disease present and no treatment administered for the last 3 years.
* Life expectancy of < 2 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-03; Primary Completion 2015-11 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Sharma, MD, Principal Investigator — University of Kansas Medical Center
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cotton-O-Neil Cancer Center (Stormont Vail Health Care), Topeka, Kansas
  - Truman Medical Center, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib: lapatinib + Endocrine therapy (will continue prior antihormone therapy, on which progression was noted)
  lapatinib: lapatinib 1500 mg PO daily
Period: Overall Study
Arm/Group | Lapatinib
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival (PFS) will be defined as the interval between the date of study initiation and the earliest date of disease progression, determined by tumor assessment.
Time Frame: 12 months
Measure: Median (80% Confidence Interval); unit: months
Groups:
- Lapatinib: lapatinib + Endocrine therapy
  lapatinib: lapatinib 1500 mg PO daily
Arm/Group | Lapatinib
Number analyzed (Participants) | 33
months | 2.1 [1 to 12]

ADVERSE EVENTS:
Time Frame: 5 years (2009-2014)
Arm/Group | Lapatinib
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 6/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (N=33)
Neck pain (General disorders) | 1
Pancreatitis (Hepatobiliary disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Skin infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Blurred vision (Eye disorders) | 1
Gait abnormal (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (N=33)
Abdominal pain (General disorders) | 2
Abducens nerve disorder (Nervous system disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 9
Acoustic nerve disorder NOS (Nervous system disorders) | 1
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1
Anorexia (Psychiatric disorders) | 7
Anxiety (Nervous system disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Auditory/Ear - Other (Specify) (Ear and labyrinth disorders) | 1 — fullness in the right ear without pain
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Bronchitis (Infections and infestations) | 1
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 1
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine increased (Metabolism and nutrition disorders) | 1
Dehydration (Gastrointestinal disorders) | 5
Depression (Psychiatric disorders) | 1
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 — scratches on back
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 — irritation at breast folds
Diarrhea (Gastrointestinal disorders) | 25
Diplopia (Eye disorders) | 1
Dizziness (Nervous system disorders) | 4
Dry mouth (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 — mouth sores/ulcerations
Edema limbs (General disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 10
Fecal incontinence (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Flu-like syndrome (General disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Gastric infection (Infections and infestations) | 1
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3
Headache (General disorders) | 6
Hearing (without monitoring program) (Ear and labyrinth disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Endocrine disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Infection, Upper airway NOS (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 4
Joint pain (Musculoskeletal and connective tissue disorders) | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 1
Memory impairment (Psychiatric disorders) | 1
Mucosal infection (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nasal/paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neurology - Other (Specify) (Nervous system disorders) | 1 — feet feel hot but no fever
Neutrophils low (Blood and lymphatic system disorders) | 2
Ocular - Other (Specify) (Eye disorders) | 1 — left eye ptosis
Oral pain (Gastrointestinal disorders) | 2
Pain in extremity (General disorders) | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 12
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Rigors/chills (General disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Vasovagal episode (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Weight loss (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No